CLINICAL TRIAL: NCT00426881
Title: The Effect of Resistance Training on Cognitive Performance, Cortical Plasticity, and Fall Risk in Women Aged 65-75 Years Old: A 12-Month RCT
Brief Title: Brain Power: Resistance Training and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Michael Smith Foundation for Health Research (Other)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: H06-03216; ORSIL 06-1737; ORSIL 05-6933
Record Dates: First submitted 2007-01-23; First posted 2007-01-25 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: Exercise; Resistance training
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Twice weekly resistance training for 52 weeks.
  Interventions: Behavioral: Exercise Training
- 2 (Experimental): Once weekly resistance training for 52 weeks.
  Interventions: Behavioral: Exercise training
- 3 (Experimental): Twice weekly balance and tone training for 52 weeks.
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise Training — Twice weekly resistance training for 52 weeks.
  Arms: 1
Behavioral: Exercise training — Once weekly resistance training for 52 weeks.
  Arms: 2
Behavioral: Exercise training — Twice weekly resistance training for 52 weeks.
  Arms: 3

SUMMARY:
Primary Objectives:

1. To ascertain whether a 12-month, twice-weekly or once-weekly resistance training (RT) program will significantly improve executive function in community-dwelling women aged 65 to 75 years old compared with a 12-month, twice-weekly stretch and relax (S & R) program (shame exercise). We will assess executive function by standard neuropsychological tests.

Secondary Objectives:

1. To describe the neural mechanisms that underpin the observed changes in executive function associated with a 12-month, twice-weekly or once-weekly RT training (by using functional magnetic resonance imaging (fMRI)).
2. To investigate whether RT-induced changes in executive function are independently associated with changes in physiological fall risk profile.
3. To investigate the dose response of RT (resistance training) on bone health as measured by dual energy x-ray and peripheral quantitative computed tomography.
4. To conduct a one-year follow-up after the formal cessation of the resistance training programs to determine the persisting effect of resistance training on cognitive performance, cortical plasticity, physiological falls risk, and bone health.

DETAILED DESCRIPTION:
Primary Research Question: Does resistance training (RT) significantly improve cognitive function, specifically executive function in older women with a Mini-Mental State Examination (MMSE) score equal to or greater than 24 (i.e., cognitively intact) compared with a stretch & relax (S & R; control) program?

Secondary Research Questions:

1. Are changes in cortical activation associated with RT-induced changes in executive function?
2. Are RT-induced improvements in executive function associated with lowered physiological fall risk?
3. Is there a dose-response on bone health with RT (resistance training)?

RESEARCH PLAN:

Study Design: A 12-month, single-blinded, randomized controlled trial. Participants: 155 cognitively-intact (i.e., MMSE score > 24), right-handed, sedentary community-dwelling women, aged 65 to 75 years.

Measurement: Measurements will take place at baseline, six month, and trial completion. Standard neuropsychological testing and physiological fall risk assessment will occur at all three measurement sessions. A subset of the participants (20 from each experimental group) will undergo fMRI assessment at baseline and trial completion only. Exercise Classes: Participants will be randomized to a 12-month, twice-weekly or once-weekly RT program or stretch & relax program (control). All exercises will be offered at a Vancouver YMCA with whom we have partnered previously. Sample Size Justification: The sample size of 50 per experimental group (i.e., N = 155) is based on the primary end point of this study, cognitive performance of executive function. SUMMARY: Falls are a major challenge for the senior population. To date, no intervention has significantly reduced falls among those with cognitive impairment. Our immediate primary goal is to test whether RT can improve cognitive performance of executive function; impaired executive function are associated with injurious falls. If this proposed exercise trial proves successful, the RT intervention will be trialed in the future in a larger study powered for falls.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (less than twice weekly exercising) women aged 65-75 years old without conditions restricting them from exercising.

Ages: 65 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 155 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Cognitive Performance of Executive Function | 12 months

SECONDARY OUTCOMES:
Functional MRI and physiological falls risk | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Liu-Ambrose, Ph.D, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - YMCA, Vancouver, British Columbia
  - Vancouver Coastal Health Research Institute Research Pavilion, Vancouver, British Columbia

REFERENCES:
- [Derived] Bolandzadeh N, Tam R, Handy TC, Nagamatsu LS, Hsu CL, Davis JC, Dao E, Beattie BL, Liu-Ambrose T. Resistance Training and White Matter Lesion Progression in Older Women: Exploratory Analysis of a 12-Month Randomized Controlled Trial. J Am Geriatr Soc. 2015 Oct;63(10):2052-60. doi: 10.1111/jgs.13644. Epub 2015 Oct 12. PMID 26456233
- [Derived] Davis JC, Nagamatsu LS, Hsu CL, Beattie BL, Liu-Ambrose T. Self-efficacy is independently associated with brain volume in older women. Age Ageing. 2012 Jul;41(4):495-501. doi: 10.1093/ageing/afs029. Epub 2012 Mar 21. PMID 22436405
- [Derived] Nagamatsu LS, Hsu CL, Handy TC, Liu-Ambrose T. Functional neural correlates of reduced physiological falls risk. Behav Brain Funct. 2011 Aug 16;7:37. doi: 10.1186/1744-9081-7-37. PMID 21846395
- [Derived] Davis JC, Marra CA, Robertson MC, Najafzadeh M, Liu-Ambrose T. Sustained economic benefits of resistance training in community-dwelling senior women. J Am Geriatr Soc. 2011 Jul;59(7):1232-7. doi: 10.1111/j.1532-5415.2011.03474.x. Epub 2011 Jun 30. PMID 21718265
- [Derived] Davis JC, Marra CA, Liu-Ambrose TY. Falls-related self-efficacy is independently associated with quality-adjusted life years in older women. Age Ageing. 2011 May;40(3):340-6. doi: 10.1093/ageing/afr019. Epub 2011 Mar 24. PMID 21436152
- [Derived] Davis JC, Marra CA, Beattie BL, Robertson MC, Najafzadeh M, Graf P, Nagamatsu LS, Liu-Ambrose T. Sustained cognitive and economic benefits of resistance training among community-dwelling senior women: a 1-year follow-up study of the Brain Power study. Arch Intern Med. 2010 Dec 13;170(22):2036-8. doi: 10.1001/archinternmed.2010.462. No abstract available. PMID 21149764
- [Derived] Liu-Ambrose T, Davis JC, Nagamatsu LS, Hsu CL, Katarynych LA, Khan KM. Changes in executive functions and self-efficacy are independently associated with improved usual gait speed in older women. BMC Geriatr. 2010 May 19;10:25. doi: 10.1186/1471-2318-10-25. PMID 20482830
- [Derived] Davis JC, Marra CA, Najafzadeh M, Liu-Ambrose T. The independent contribution of executive functions to health related quality of life in older women. BMC Geriatr. 2010 Apr 1;10:16. doi: 10.1186/1471-2318-10-16. PMID 20359355
- [Derived] Liu-Ambrose T, Nagamatsu LS, Graf P, Beattie BL, Ashe MC, Handy TC. Resistance training and executive functions: a 12-month randomized controlled trial. Arch Intern Med. 2010 Jan 25;170(2):170-8. doi: 10.1001/archinternmed.2009.494. PMID 20101012